CLINICAL TRIAL: NCT07136103
Title: A First-in-Human Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of ABBV-277 in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of ABBV-277 in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: M24-934
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; ABBV-277

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (10):
- Group 1: ABBV-277-Dose A (Experimental): Participants will receive ABBV-277 Dose A on day 1 and followed for 196 days
  Interventions: Drug: ABBV-277
- Group 1: Placebo (Experimental): Participants will receive Placebo on day 1 and followed for 196 days
  Interventions: Drug: Placebo
- Group 2: ABBV-277-Dose B (Experimental): Participants will receive ABBV-277 Dose B on day 1 and followed for 196 days
  Interventions: Drug: ABBV-277
- Group 2: Placebo (Experimental): Participants will receive Placebo on day 1 and followed for 196 days
  Interventions: Drug: Placebo
- Group 3: ABBV-277-Dose C (Experimental): Participants will receive ABBV-277 Dose C on day 1 and followed for 196 days
  Interventions: Drug: ABBV-277
- Group 3: Placebo (Experimental): Participants will receive Placebo on day 1 and followed for 196 days
  Interventions: Drug: Placebo
- Group 4: ABBV-277-Dose D (Experimental): Participants will receive ABBV-277 Dose D on day 1 and followed for 196 days
  Interventions: Drug: ABBV-277
- Group 4: Placebo (Experimental): Participants will receive Placebo on day 1 and followed for 196 days
  Interventions: Drug: Placebo
- Group 5: ABBV-277-Dose E (Experimental): Participants will receive ABBV-277 Dose E on day 1 and day 2 and followed for 196 days
  Interventions: Drug: ABBV-277
- Group 5: Placebo (Experimental): Participants will receive Placebo on day 1 and day 2 and followed for 196 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABBV-277 — • Intravenous (IV) infusion
  Arms: Group 1: ABBV-277-Dose A; Group 2: ABBV-277-Dose B; Group 3: ABBV-277-Dose C; Group 4: ABBV-277-Dose D; Group 5: ABBV-277-Dose E
Drug: Placebo — • Intravenous (IV) infusion
  Arms: Group 1: Placebo; Group 2: Placebo; Group 3: Placebo; Group 4: Placebo; Group 5: Placebo

SUMMARY:
The objective of this study is to evaluate the safety, tolerability, immunogenicity and pharmacokinetics (PK ) properties following a single dose of ABBV-277 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 35 kg
* Body Mass Index (BMI) is ≥ 18.0 to ≤ 32.0 kg/m^2 after rounding to the tenths decimal.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile neurological examination, and a 12-lead ECG

Exclusion Criteria:

* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), endocrine, metabolic, renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
* Participant must meet pregnancy/conception/partner considerations criteria as detailed in the eligibility section.
* Participants using any medications, vitamins and/or herbal supplements within the 14-day period prior to study drug administration or within 5 half-lives of the respective medication, whichever is longer.
* History of any clinically significant illness/infection/major febrile illness, hospitalization, or any surgical procedure within 30 days prior to the first dose of study drug.
* History of suicidal ideation currently or within one year prior to study drug administration as evidenced by answering "yes" to Questions 4 or 5 on the suicidal ideation portion of the C - SSRS completed at screening, or any history of suicide attempts within the last two years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of ABBV-277 | Up to approximately 9 days
  Cmax of ABBV-277
Time to Cmax (Tmax) of ABBV-277 | Up to approximately 9 days
  Tmax of ABBV-277
Terminal Phase Elimination Rate Constant (Beta) of ABBV-277 | Up to approximately 9 days
  Terminal phase elimination rate constant (beta) of ABBV-277
Terminal Phase Elimination Half-Life (t1/2) of ABBV-277 | Up to approximately 9 days
  Terminal phase elimination half-life of ABBV-277
Area Under the Concentration-Time Curve From Time 0 to Time t (AUCt) of ABBV-277 | Up to approximately 9 days
  AUCt of ABBV-277
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of ABBV-277 | Up to approximately 9 days
  AUCinf of ABBV-277
Number of Participants With Adverse Events (AEs) | Up to Day 196
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 265681, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-934